CLINICAL TRIAL: NCT04760132
Title: National Cohort Study of Effectiveness and Safety of SARS-CoV-2/COVID-19 Vaccines
Brief Title: National Cohort Study of Effectiveness and Safety of SARS-CoV-2/COVID-19 Vaccines (ENFORCE)
Acronym: ENFORCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jens D Lundgren, MD (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Sponsor-Investigator, Jens D Lundgren, MD, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ENFORCE
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV Infection
Keywords: COVID-19; Vaccination
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Injections

STUDY DESIGN:
Intervention Model Description: The design is an open-labelled, non-randomised, parallel group, phase IV study with historical controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccine A - COMIRNATY COVID-19 vaccine (Active Comparator): COMIRNATY (COVID-19, mRNA Vaccine) by BioNTech Manufacturing GmbH Marketing Authorisation EU/1/20/1528
  Interventions: Biological: COMIRNATY - BioNTech Manufacturing GmbH
- Vaccine B - Moderna COVID-19 vaccine (Active Comparator): COVID-19 Vaccine Moderna dispersion for injection (COVID-19, mRNA Vaccine) by MODERNA BIOTECH SPAIN S.L.
  Marketing Authorisation EU/1/20/1507/001
  Interventions: Biological: COVID-19 Vaccine Moderna dispersion for injection - MODERNA BIOTECH
- Vaccine C - Astra-Zeneca COVID-19 vaccine (Active Comparator): COVID-19 Vaccine AstraZeneca suspension for injection (ChAdOx1-S [recombinant]) by AstraZeneca AB Marketing Authorisation EU/1/21/1529/001 and /002
  Interventions: Biological: COVID-19 Vaccine AstraZeneca suspension for injection

INTERVENTIONS:
Biological: COMIRNATY - BioNTech Manufacturing GmbH — Vaccination as part of the the Danish national government programme
  Arms: Vaccine A - COMIRNATY COVID-19 vaccine
Biological: COVID-19 Vaccine Moderna dispersion for injection - MODERNA BIOTECH — Vaccination as part of the the Danish national government programme
  Arms: Vaccine B - Moderna COVID-19 vaccine
Biological: COVID-19 Vaccine AstraZeneca suspension for injection — Vaccination as part of the the Danish national government programme
  Arms: Vaccine C - Astra-Zeneca COVID-19 vaccine

SUMMARY:
National cohort study of effectiveness and safety of SARS-CoV-2 vaccines (ENFORCE is an equivalence trial to evaluate the effectiveness and safety of multiple new SARS-CoV-2 vaccines approved for use in the EU, and which are being offered at participating units.

The design is an open-labelled, non-randomised, parallel group, phase IV study with historical controls.

A sub-study will be embedded within this master protocol addressing basic and translational research questions requiring additional sampling of biological material (under separate participant informed consent).

DETAILED DESCRIPTION:
First phase will enrol 10,000 persons initiating vaccination (assuming 4 vaccines). If more vaccines become available additional 2,500 persons per vaccine will be included. Subsequent phases with larger sections of the population included may be implemented.

Participants will have 6 study visits and be followed for 2 years after the first vaccination, which offers the participants an extra close follow up on vaccine effectiveness. Safety data will be collected at study visits until 3 months after the first vaccination. Research samples will be collected at each study visit during the two year follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related procedures are performed
2. Male or female eligible for SARS-CoV-2 immunization (as defined by SST in the national vaccination plan)
3. The subject must be willing and able to comply with trial protocol (re-visits and biological samples)

Exclusion Criteria:

1. Male and female under the age of 18
2. Any subgroup of individuals for which the vaccines are contraindicated
3. Previous SARS-CoV-2 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7600 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the effectiveness of citizens being vaccinated with one of the SARS-CoV-2 vaccines | The change from Base-line in MPNAT measured via profiling of antibodies against SARS-CoV-2 Spike epitopes at 24 month
  Primary outcome is the minimal protective neutralising antibody titre (MPNAT); i.e. the minimum level of neutralising antibodies sufficient to protect the person from becoming infected.

SECONDARY OUTCOMES:
Number of breakthrough infections in the 24 months period will be used to compare the effectiveness between the vaccines | The change from first vaccination until 24 month
  Number of confirmed positive SARS-CoV-2 tests reported via the national testing system.
Assessment of the safety of the vaccines will be compared between groups | From first vaccine until Day 90
  Reports of participants with local and systemic reactions to the vaccination will be collected
Assessment of any Adverse Event from the vaccines will be compared between groups | From first vaccine until Day 90
  Reports of participants with grade 3 and 4 Adverse Events and any Serious Adverse will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Professor, Study Chair — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Aarhus Universitetshospital, Skejby, Aarhus, Aarhus N
  - Aalborg Universityhospital Syd, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Odense Universityhospital, Odense
  - Sjællandsuniversitetshospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staerke NB, Reekie J, Johansen IS, Nielsen H, Benfield T, Wiese L, Sogaard OS, Tolstrup M, Iversen KK, Tarp B, Larsen FD, Larsen L, Lindvig SO, Holden IK, Iversen MB, Knudsen LS, Fogh K, Jakobsen ML, Traytel AK, Ostergaard L, Lundgren J; ENFORCE Study Group. Cohort Profile:The Danish National Cohort Study of Effectiveness and Safety of SARS-CoV-2 vaccines (ENFORCE). BMJ Open. 2022 Dec 30;12(12):e069065. doi: 10.1136/bmjopen-2022-069065. PMID 36585137